CLINICAL TRIAL: NCT06853262
Title: Influence of Manual Therapy on the Motor and Non-motor Symptoms of Parkinson's Disease
Brief Title: Manual Therapy in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Juan Elicio Hernández Xumet, Principal Investigator; Clinical Professor; Head of the Clinical Research Laboratory - Physiotherapy Department, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUC_2024_28
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Therapy Protocol (Experimental): The study subjects will receive a maximum of two manual therapy sessions per week for a minimum of six weeks. The variables will be measured before and after the six weeks for the secondary variables and during all the sessions for the main variables of nervous system activity.
  The intervention protocol consists of a maximum of 15 manual therapy techniques, which will always be carried out in the same order. The estimated time for each technique is 90 seconds. Therefore, the intervention protocol will last approximately 25-35 minutes.
  Before starting treatment, the patient will receive a document with all the information regarding the study and the informed consent form, which the research team must fill out and sign before the intervention.
  Interventions: Other: Manual Therapy Protocol
- Sham Manual Protocol (Sham Comparator): Manual intervention protocol with placebo techniques where the hands are placed on the same areas as in the experimental protocol techniques
  Interventions: Other: Sham Manual Protocol

INTERVENTIONS:
Other: Manual Therapy Protocol — The techniques were divided into three main groups: first, those carried out in transverse planes, then carried out in a specific zone, and finally, those aimed at the course of the vagus nerve. The techniques are carried out by physiotherapists with more than 15 years of healthcare experience and trained in manual therapy with more than 10 years of experience in this field.
  Arms: Manual Therapy Protocol
Other: Sham Manual Protocol — The Sham techniques were divided into three main groups: first, those carried out in transverse planes, then carried out in a specific zone, and finally, those aimed at the course of the vagus nerve. The Sham techniques are carried out by physiotherapists with more than 15 years of healthcare experience and trained in manual therapy with more than 10 years of experience in this field.
  Arms: Sham Manual Protocol

SUMMARY:
An experimental study will be carried out to examine how a manual therapy protocol can influence a series of parameters related to motor and non-motor symptoms in patients who have Parkinson's disease / Parkinsonism.

To do this, an intervention will be carried out that will last a minimum of 6 weeks. In addition to their ongoing treatment, the study subjects will receive a maximum of 2 sessions of manual therapy each week. They will undergo a series of measurements both before and after the intervention related to gait, balance, non-motor symptoms, and some more specific parameters of gait.

The study's main objective is to obtain information about possible treatment models based on manual therapy for Parkinson's disease. It is also hoped to compile a series of results that will lead to conclusions and benefit the development of physiotherapy for this disease. It is also hoped that this will help those affected so that the treatment is as comprehensive as possible and that the physiotherapist can use as many tools as are available to them to address the pathology.

ELIGIBILITY:
Inclusion Criteria:

* People aged between 40 and 75 who voluntarily agree to take part in this study

Exclusion Criteria:

* People with Dementia and established cognitive impairment with scores on the Montreal Cognitive Assessment Test (MoCA) of less than 25

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Autonomic nervous system activity | Baseline and every six weeks for up to 6 months from the start
  To evaluate the activity of the ANS through the indices of the Sympathetic Nervous System (SNS) and Parasympathetic Nervous System (PNS). These two parameters are the main variables of the study and were evaluated before, during and after the manual protocols to be applied. For this purpose, the Elite HRV smartphone application was used, which connects to a Polar transmitter band placed on the person's chest at the level of the xiphoid process of the sternum, which allowed constant monitoring of the subject during each of the interventions.

SECONDARY OUTCOMES:
PD NMS Quest | Baseline and every six weeks for up to 6 months from the start
  PD NMS Quest: this is the questionnaire for non-motor symptoms in Parkinson's disease. It consists of 30 yes or no questions.
Mini-BESTest | Baseline and every six weeks for up to 6 months from the start
  Mini-BESTest: identified as the most comprehensive balance measurement for adults and the elderly. It has a series of items with their corresponding score, the maximum score that can be obtained at the end of the test is 28 points.
Berg Balance Scale | Baseline and every six weeks for up to 6 months from the start
  Berg Balance Scale: allows the static and dynamic balance abilities of a person to be assessed. Like other tests and scales, it has a series of items and the maximum score that can be achieved at the end of the test is 56 points.
Timed Up and Go (TUG) | Baseline and every six weeks for up to 6 months from the start
  Timed Up and Go (TUG): this is a test that consists of getting up from a chair, walking to a mark 3 metres away, turning around and sitting back down in the same chair. The time taken to complete the test is measured.
Tinetti scale | Baseline and every six weeks for up to 6 months from the start
  Tinetti scale: used to detect the risk of falls in the elderly, it consists of a series of items with their corresponding score. The maximum score that can be obtained at the end of the test is 28 points.
Range of Motion (ROMs) | Baseline and every six weeks for up to 6 months from the start
  Range of Motion (ROMs): using slow-motion recordings from a sagittal plane, the ranges of hip, knee, plantar and dorsal ankle flexion are measured while the person walks in a straight line. The recordings are then imported into software where the corresponding analyses of the captured images are carried out. The results are expressed in degrees.
Walk Measure | Baseline and every six weeks for up to 6 months from the start
  Stride length: the distance between the points of contact of the alternating feet with the ground. To evaluate this variable, the same process is used as for the ROMs (using slow-motion videos and subsequent analysis). The results are expressed in centimetres (cm).
  Bipodal support time: this is the time that both feet are supported on the ground while walking. To evaluate this variable, the same process was carried out as with the ROMs and the length of the step (using slow motion videos and subsequent analysis). The results are expressed in milliseconds (ms).
  Stride time: this is the time interval between two successive contacts of the same foot on the ground. To evaluate this variable, the same process is used as for ROMs, stride length and bipodal support time (using slow motion videos and subsequent analysis). The results are expressed in milliseconds (ms).

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ciencias de la Salud, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No